CLINICAL TRIAL: NCT04756570
Title: The Effect of Robot-Assisted Gait Training Dose on Walking, Functional Recovery and Quality of Life in Stroke Patients
Brief Title: The Effect of Robot-Assisted Gait Training in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Physical Med-3
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Stroke
Keywords: Rehabilitation; Robotic; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Three groups with one control group
Who Masked: Outcomes Assessor
Masking Description: Participant will be evaluated by an another investigator who does not aware of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): 25 stroke patients between the ages of 18-80, stroke duration of less than 2 months and not more than 2 years whose Mini-Mental State Examination (MMSE) scores equal or above the 25 will be included in this study. Modified Ashworth Scale (MAS), Barthel Index, The Modified Rankin Scale, Berg Balance Scale , &-min walk test, and Stroke-Specific Quality of Life Scale (SSQOL) assessments will be applied just before the rehabilitation program, after the application and at the end of 6 weeks
  Interventions: Other: Control
- Robotic 1 (Active Comparator): 25 stroke patients between the ages of 18-80, stroke duration of less than 2 months and not more than 2 years whose MMSE scores equal or above the 25 will be included in this study. Modified Ashworth Scale (MAS), Barthel Index, The Modified Rankin Scale, Berg Balance Scale , &-min walk test, and Stroke-Specific Quality of Life Scale assessments will be applied just before the rehabilitation program, after the application and at the end of 6 weeks
  Interventions: Other: Robotic Group 1
- Robotic 2 (Active Comparator): 25 stroke patients between the ages of 18-80, stroke duration of less than 2 months and not more than 2 years whose MMSE scores equal or above the 25 will be included in this study. Modified Ashworth Scale (MAS), Barthel Index, The Modified Rankin Scale, Berg Balance Scale , &-min walk test, and Stroke-Specific Quality of Life Scale assessments will be applied just before the rehabilitation program, after the application and at the end of 6 weeks
  Interventions: Other: Robotic Group 2

INTERVENTIONS:
Other: Control — Individuals in this group will be randomly recruited from hospitalized stroke volunteers. Since these individuals receive routine rehabilitation 5 days a week, they will be evaluated at the beginning and end of 18 sessions over a total period of 6 weeks. Conventional physiotherapy will include normal joint movements, muscle strengthening exercises, balance and mobility exercises, and exercises to improve daily life activity.
  Other Names: Conventional therapy
  Arms: Control
Other: Robotic Group 1 — Individuals in this group will receive one session of robotic rehabilitation in addition to conventional therapy each week
  Arms: Robotic 1
Other: Robotic Group 2 — Individuals in this group will receive two sessions of robotic rehabilitation in addition to conventional therapy each week
  Arms: Robotic 2

SUMMARY:
Stroke has been defined by the World Health Organization as a condition with rapid onset and vascular origin, leading to a focal or global deterioration in brain functions lasting 1 day or longer. Stroke is an important health problem affecting a large part of the society with its high frequency and mortality. Post-stroke disability reduces the patient's quality of life and causes socioeconomic and social problems. Post-stroke hemiplegia often causes a decrease in the ambulatory ability of the patient. As a result, the patient's independence to move inside and outside the home is negatively affected. Gait is one of the most affected sensorimotor functions in stroke patients. Although the majority of patients strive to walk independently, they cannot reach a level of independent walking sufficient to perform activities of daily living (ADL). Current studies emphasize that the intensive early rehabilitation program is effective in treating patients with gait and movement disorders. Rehabilitation programs with a multidisciplinary approach are the most effective options that can be applied to increase a patient's functional status and post-stroke independence. Robotic-assisted walking devices are one of the current and effective methods used to regain ambulation.

DETAILED DESCRIPTION:
Robotic-assisted walking devices are used in the treatment of many neurological diseases such as spinal cord trauma, multiple sclerosis, post-stroke hemiplegia. In treatments applied with robotic walking devices, since accurate and equal weight transfer is provided in both lower extremities, sensorimotor learning of the patient is also supported. Thanks to the intense and repetitive simulation provided in every phase of the walk and the proprioceptive inputs taken, reorganization occurs in the cortical and sub-cortical regions. With the continuous facilitation of the walking cycle, neural transmission is regenerated or existing communication is strengthened between the motor areas of the brain and sensory pathways. The advantages of robotic systems can be listed as enabling longer and more intense treatments, ensuring that the patient feels better cognitively, adapting to exercise better, providing the opportunity to check the patient's condition objectively by monitoring and recording the patient's condition functionally. A recent systematic review showed that individuals with stroke who received robotic gait training combine with physiotherapy were more likely to achieve independent walking than those who received gait training without robotic gait training. Different studies on the effectiveness of robotic rehabilitation have reported that robot-assisted gait training should be applied together with a physiotherapy program. However, there is no clear information on the optimal dosage of Robot-Assisted Gait Training (RAGT) to achieve clinically meaningful functional recovery after a central nervous system injury. This study aims to investigate the effect of RAGT dosage on Functional Recovery and Quality of Life in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stroke
* Willing to participate
* Modified Ashworth Scale Score lower than "3"
* Able to walk 10 meter independently

Exclusion Criteria:

* Secondary neurological diseases
* Cognitive problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Six weeks
  It is a scale that includes fourteen balance activities and scores between 0-4 by observing the patient's performance for each activity. This scale includes activities such as moving from a sitting position to a standing position, turning while standing, picking up objects while standing, rotating 360 degrees, standing on one foot. If the patient cannot do the activity, 0 points are given, and 4 points are given if the patient does the activity independently. Low scores indicate impaired balance. The highest total score is 56 and 0-20 points indicate an imbalance, 21-40 points indicate an acceptable balance, 41-56 points indicate the presence of a good balance.

SECONDARY OUTCOMES:
The Barthel Index | Six weeks
  The Barthel Index (BI) evaluates physical independence in activities of daily living in 10 items (transfer, ambulation / wheelchair use, climbing up and downstairs, feeding, dressing, self-care, bathing, toilet use, urinary continence, stool continence). Each item is scored separately as 0, 5, 10 or 15 points. The total score between 0-20 means fully dependent, 21-61 highly dependent, 62-90 moderately dependent, 91-99 mildly dependent and 100 fully independent. In our study, the version of the BI, which has been adapted to Turkish and whose validity and reliability study has been made, will be used.
Stroke-Specific Quality of Life Scale | Six weeks
  Stroke-Specific Quality of Life Scale was used to assess the quality of life. SSQOL consists of 12 sub-sections including energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper limb function, vision, and work productivity and a total of 49 questions. It is graded with Likert type scoring ranging from 1 to 5. It was adapted to Turkish in 2009 by Hakverdioğlu et al. A question was removed from the original scale and the subsections were grouped under 8 headings. These subheadings are; activities, social and family roles, language, vision, energy, temperament, personality and thinking.
6-min walk test | Six weeks
  6-min walk test is based on the patient walking for 6 minutes in a certain length of the corridor. Before, the patient is rested on a chair for 15 minutes. Patients are asked to walk as fast as possible at their walking speed for 6 minutes in a 30-meter straight corridor and the distance traveled is recorded.
Modified Rankin Scale | Six weeks
  The Modified Rankin Scale (MRS) is used to evaluate the disability level of individuals after stroke. Points between 0 and 6 can be obtained. 0 points indicate no symptoms, 5 points indicate bedridden and continuous care, and 6 points indicate death.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Fatih Yaşar, MD, Principal Investigator — Bolu Abant Izzet Baylsa University
Locations (1):
- Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No